CLINICAL TRIAL: NCT05308108
Title: Study of Postoperative Respiratory Complications in Children With Obstructive Sleep Apnea.
Brief Title: Study of Postoperative Respiratory Complications in Children With Obstructive Sleep Apnea (PORC)
Acronym: PORC
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Vera Saldien, Principle Investigator, University Hospital, Antwerp
Other Study IDs: 002364
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Child, Only; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Obstructive Sleepapnea
  Interventions: Procedure: (Adeno)tonsillectomy

INTERVENTIONS:
Procedure: (Adeno)tonsillectomy — registration of PORC in children with OSAS after (adeno)tonsillectomy

SUMMARY:
Adenotonsillectomy is the first line surgical treatment for children with Obstructive Sleep apnea Syndrome (OSAS). Postoperative respiratory complications (PORC) may occur and are often related to co-morbidities. Despite guidelines from different scientific groups, there is no consensus on the monitoring requirements and management of PORC in these children.

DETAILED DESCRIPTION:
Postoperative respiratory complications (PORC) may occur in children with obstructive sleep apnea undergoing upper airway surgery. The incidence of these postoperative respiratory complications can be affected by co-morbidities such as obesity, Down-syndrome, neurologic conditions, craniofacial malformation. Despite treatment guidelines from different scientific groups such as 'American Academy of Pediatrics', the 'European Respiratory Society' , the American Academy of Otorhinolaryngology and the American society of Anesthesiology, there is no consensus on the monitoring requirements and management of PORC in these children.

Further studies are required to investigate the role of age and OSAS severity on the occurence of PORC. Secondly, it would be interesting to develop a flowchart for the postoperative management of children with OSAS undergoing upper airway surgery, taking into account child-related factors such as age, OSAS and comorbidity.

As standard of care, all children are seen at the preoperative outpatient clinic by an anesthesiologist. If necessary, additional tests are performed with respect to the health condition of the child.

If all inclusion criteria are fulfilled and there are no exclusion criteria, Informed Consent will be asked of the accompanying parent or legal guardian.

Premedication is typically not indicated by these interventions because they are of short duration. In exceptional situations (for example an extremely anxious child) the use of premedication can be considered. In such a case, one can choose either midazolam sirup (Ozalin 0.25milligrams/kilogram (mg/kg) for children, 1 year or older, with a body weight of 3 to 40 kg) or Lorazepam sublingually (Temesta expidet) from an age of 6 years, dosage 0.5 mg for body weight of 25-50kg and dosage of 1 mg for body weight of 50 kg and more).

Per-operative anesthetic management: basic monitoring includes Electrocardiogram, non-invasive blood pressure monitoring, pulse oximetry, end-tidal carbon dioxide (EtCO2) and body temperature, intravenous (IV) access with administration of IV fluids as per body weight as standard of care. At the start of the intervention, venous access is obtained during inhalational anesthesia.

Drug-induced sleep endoscopy (DISE) is performed with IV propofol and/or sevoflurane. Induction of anesthesia occurs with IV propofol or inhalational anesthesia with sevoflurane. If propofol IV is used, a bolus of 10-20 mg and continuous infusion 6-10 mg/kg/hr is administered.

After the DISE examination, the child is intubated with fentanyl 2 micrograms/kg or sufentanil 0.2 micrograms/kg according to the clinical presentation. For neuromuscular block, atracurium 0.2 to 0.3 mg per kg is used. For maintenance of anesthesia a minimum alveolar concentration (MAC) 1 to 1.5 sevoflurane is kept.

Postoperative pain management is achieved by a combination of analgesics (non-steroidal anti-inflammatory drugs and paracetamol) as per age-specific indications (IV paracetamol 20mg/kg, ketorolac 0.5 mg/kg and morfine 0.05 mg/kg in cases of tonsillectomy) Postoperative nausea and vomiting is prevented by a single shot dexamethasone 0.15 milligram/kilogram IV.

After surgery, when the patient is awake he or she will be extubated and transferred to the Post Anesthetic Care Unit (PACU or recovery room) for monitoring of vital signs. Minimal requirement in the recovery room is a peripheral saturation monitor.

Monitoring of postoperative respiratory complications starts at end of surgery. So if a child develops respiratory problems upon awakening from anesthesia but before admission to the recovery room, these will also be registered as postoperative respiratory complications. Possible PORC are: laryngospasm, bronchospasm, desaturation requiring Oxygen, pulmonary edema.

In case of occurrence of PORC, the following interventions will be applied per protocol:

* oxygen saturation level between 92-95%: adopt lateral position
* oxygen saturation below 92% : administer oxygen (O2) via nasal prongs 1 Liter/ Minute (L/M)
* monitoring pulse oximetry for 2 minutes;
* in case of no response, increase O2 therapy via nasal prongs to 1.5 L/M
* monitoring pulse oximetry for 2 minutes;
* in case of no response, O2 therapy via nasal prongs will be increased to 2 L/M
* monitoring pulse oximetry for 2 minutes
* in case of no response, increase O2 therapy via nasal prongs to 2.5 L/M
* monitoring pulse oximetry for 2 minutes
* in case of no response, increase O2 therapy via nasal prongs to 3 L/M
* monitoring pulse oximetry for 2 minutes
* in case of no response, increase O2 therapy via nasal prongs to 3.5 L/M
* monitoring pulse oximetry for 2 minutes
* in case of no response, increase O2 therapy via nasal prongs to 4 L/M
* If pulse oximetry stays below 92 % despite standard O2 therapy at 4 L/M, nasal high flow therapy (Optiflow) will be applied according to the bodyweight.
* Flow = 2 l/kg/min with fraction of inspired oxygen (FiO2) 50% for bodyweight up to 10kg. If bodyweight > 10 kg add 0.5 l/kg/min extra
* monitor for 2 minutes
* If no improvement, Optiflow with FIO2 80%
* In case of persistent low pulse oximetry (below 92%) and no improvement of clinical symptoms, patient will be intubated and transferred to the Pediatric Intensive Care Unit (PICU)
* Postoperative pain management during first 24H after surgery: Paracetamol 15 mg/kg 4 times a day and Taradyl 0.5 mg/kg 3 times/day
* PORC will be registered every 30 minutes the first 6H postoperative. Upon arrival at the ward, PORC will be registered for 24 hours.
* All patients stay at least one night in hospital for overnight pulse oximetry monitoring

When the clinical parameters are stable for 30 minutes, at any time of the study protocol, the registration period for the study ends. Further management according to the responsible physician.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for (adeno)tonsillectomy as treatment for OSAS

Exclusion Criteria:

* other surgery than (adeno)tonsillectomy performed as treatment for OSAS
* Polysomnography not available within 1 year before surgery

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with or without co-morbidities undergoing (adeno)tonsillectomy for OSAS during time frame of the study period
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
The incidence of PORC related to age in children with/without comorbidities undergoing (adeno)tonsillectomy | 24hr postoperative period
  Number of PORC
The incidence of PORC related to OSAS severity in children with/without comorbidities undergoing (adeno)tonsillectomy | 24 hr postoperative period
  Number of PORC

SECONDARY OUTCOMES:
Development of a flow chart for postoperative monitoring of PORC in children with OSA | 2 years
  Flowchart

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD,PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium